CLINICAL TRIAL: NCT02661269
Title: Relation Between the Increase of Peripheral Edema by Fluid Therapy and the Decrease in Microcirculatory Vesseldensity
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Gerke Veenstra, MD, Frisius Medisch Centrum
Other Study IDs: nWMO 127
Record Dates: First submitted 2015-12-02; First posted 2016-01-22 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2017-03

CONDITIONS: Edema; Sepsis
MeSH Terms: conditions — Edema; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Septic patients: Septic patients with fluid overload (fluid balance + 4 L)
  Interventions: Device: Videomicroscopy of the sublingual microcirculation; Device: Bio-impedance measurements.
- Post-cardiac surgery patients: Patients after cardiac surgery, at arrival on ICU.
  Interventions: Device: Videomicroscopy of the sublingual microcirculation; Device: Bio-impedance measurements.

INTERVENTIONS:
Device: Videomicroscopy of the sublingual microcirculation — Measuring total vessel density with the Cytocam-IDF camera.
Device: Bio-impedance measurements. — measuring resistance and reactance with the BIVA method.

SUMMARY:
Can videomicroscopy of the sublingual microcirculation detect the increase in edema before peripheral edema will appear? By measuring the decrease in vesseldensity after strong positive fluid balances within septic patients versus euvolemic post-cardiac surgery patients. Measuring reactance and resistance (BIVA method) to determine volume status.

Primary outcome:

- Total vessel density (TVD)

Secondary outcome:

* Fluid balance
* BIVA measurements (reactance & resistance)

DETAILED DESCRIPTION:
There are a lot of methods to determine if a patient is fluid-responsive, however a moment to stop fluid therapy is lacking. So the purpose of this study is to find a 'stop' moment for fluid therapy before peripheral edema will be present.

With sublingual measurements of the vessel density with the Cytocam-IDF, comparing the septic patients with fluid overload , euvolemic post-cardiac surgery patients at the arrival on the ICU and healthy volunteers we can determine if there is a decrease in vessel density during fluid loading.

To give a accurate view on fluid overload we include a bio-impedance measurement of reactance and resistance. Fluid balances are recorded very accurate by our electronic patient record.

ELIGIBILITY:
Inclusion Criteria:

* after cardiac surgery
* septic patient with a fluid balance of 4L +

Exclusion Criteria:

* recent maxillofacial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU population
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Difference in vessel density (mm/mm2) of the sublingual microcirculation between the two groups. | Cardiac surgery within 4 hours of ICU admittance, 1 offline total vessel density measurement, Septic patients +/- third day of ICU admittance, 1 offline total vessel density measurement.
  With the Cytocam-IDF we make movies off the sublingual microcirculation for 6 seconds on 3 different spots, with offline analysis we calculate a mean total vessel density (total surface of vessels divided by total area surface).
  The cardiac surgery group will be measured within 4 hours of admittance on the ICU. The septic patients group will be measured on the moment that the highest fluid balance during the ICU stay, so on the moment that there will be started with diuretics of renal replacement therapy to induce a negative fluid balance.

SECONDARY OUTCOMES:
The correlation between a increasing fluid balance and the total vessel density in both groups separately. | The cumulative fluidbalance (L) will be noted at the same moment as the microcirculation movies are made, this will be the cumulative fluid balance as measured on the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: E.C. Boerma, MD-PhD, Principal Investigator — Frisius Medisch Centrum
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands